CLINICAL TRIAL: NCT06652035
Title: Possible Pharmacological Effect of Quercetin in the Management of Hyperuricemia
Brief Title: Possible Pharmacological Effect of Quercetin in the Management of Hyperuricemia - Results From Real-life Clinical Studies
Status: Completed | Type: Observational
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: The University of Urbino Carlo Bo, Italy (Unknown)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Other Study IDs: 88_18.01.2023_QuercetinFit - A
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supplemental Quercetin group: These participants received oral 500 mg Quevir® (Quercetin Phytosome®) tablet, twice a day for 90 days. Each Quevir® tablet contains 200 mg pure Quercetin.
  Interventions: Dietary Supplement: Quevir® (Quercetin Phytosome®)
- Supplemental Probiotic Strptococcus salivarius K12 (ATCC BAA-1024) group: These participants received orally dissolving Bactoblis® tablet, once daily before bedtime for 90 days. Each Bactoblis® tablet contains at least 1x10⁹ CFU of probiotic S. salivarius K12 (ATCC BAA-1024).
  Interventions: Dietary Supplement: Bactoblis®

INTERVENTIONS:
Dietary Supplement: Quevir® (Quercetin Phytosome®) — 500 mg Quevir® (Quercetin Phytosome®) tablet
  Other Names: Quevir®
  Groups: Supplemental Quercetin group
Dietary Supplement: Bactoblis® — Probiotic Streptococcus Salivarius K12 (ATCC BAA-1024)
  Groups: Supplemental Probiotic Strptococcus salivarius K12 (ATCC BAA-1024) group

SUMMARY:
Quercetin, a natural flavonoid found in various fruits and vegetables, has gained attention for its potential role in managing hyperuricemia. Emerging evidence suggests that quercetin may reduce plasma uric acid levels by inhibiting xanthine oxidase, an enzyme responsible for uric acid production. Additionally, its anti-inflammatory and antioxidant properties could help mitigate the oxidative stress and inflammation associated with hyperuricemia. As a result, quercetin supplementation offers a promising avenue for therapeutic intervention in conditions like gout and other uric acid-related disorders.

DETAILED DESCRIPTION:
In the present retrospective cross-sectional observational study, the investigators assessed the potential pharmacological effect of supplemental quercetin on the plasma uric acid levels of health adults. These participants visited nutritional clinics in Italy during the Coronavirus disease (COVID-19) pandemic for general health check-up in real-life to enhance their immune system with supplements aimed at providing additional protection against COVID-19 infection. The supplements, either quercetin or probiotic Streptococcus salivarius K12 (BLIS K12), were advised randomly to the participants for 90 days, tailored to individual needs and in the absence of any pre-defined criteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* BMI between 18.5 and 29.9 kg/m²
* Non-smoker
* Consumtion of less than 3 units of alcohol per day

Exclusion Criteria:

* - Plasma uric acid concentrations above 7 mg/dL
* Diagnosis of endocrinological, metabolic, oncological, neurological, or bowel inflammatory disease diseases, gout, kidney stones

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants visited the nutritional clinics during the COVID-19 pandemic for general health check up to improve their immunological protection against COVID-19 infection.
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in plasma uric acid level | 90 days
  Supplement effect on plasma uric acid level

SECONDARY OUTCOMES:
Change in plasma cholesterol level | 90 days
  Supplement effect on plasma cholesterol level
Change in plasma triglycerides level | 90 days
  Supplement effect on plasma triglycerides level
Change in plasma glucose level | 90 days
  Supplement effect on plasma glucose level
Change in plasma insulin level | 90 days
  Supplement effect on plasma insulin level
Change in plasma creatine phosphokinase level | 90 days
  Supplement effect on plasma creatine phosphokinase level
Change in alanine transaminase level | 90 days
  Supplement effect on liver function
Change in aspartate aminotransferase level | 90 days
  Supplement effect on liver function
Change in alkaline phosphatase level | 90 days
  Supplement effect on liver function
Change in gamma-glutamyl transferase level | 90 days
  Supplement effect on liver function
Change in bilirubin level | 90 days
  Supplement effect on liver function
Incidence of side effects | 90 days
  Number of patients reporting side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Buccomino Medical Clinic, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Pierro F, Rabbani F, Tareen M, Nigar R, Khan A, Zerbinati N, Tanda ML, Cazzaniga M, Bertuccioli A, Falasca P, Damiani G, Villanova N. Potential pharmacological effect of Quercetin Phytosome in the management of hyperuricemia: results from real-life clinical studies. Front Nutr. 2025 Feb 7;12:1519459. doi: 10.3389/fnut.2025.1519459. eCollection 2025. PMID 39990611